CLINICAL TRIAL: NCT03124563
Title: Planning the Next Steps: Using an Implementation Intention Approach to Increase Daily Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandeis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WalkingIntentions #15147
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-07

CONDITIONS: Sedentary Lifestyle; Self Efficacy; Control Locus
Keywords: Exercise; Health Behavior; Aging
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Health Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants are aware of the nature of the intervention. They are not aware if they are the experimental or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Participants will wear a Fitbit Zip to record their daily activity data, which will be deidentified and aggregated with an online platform called Fitabase. Participants in the control group will be matched with the intervention group for how much contact they have with the researcher.
  Interventions: Behavioral: Control Group
- Implementation Intention Condition (Experimental): Participants will wear a Fitbit Zip to record their daily activity data, which will be deidentified and aggregated with an online platform called Fitabase. Participants in this arm will receive all components of the intervention: scheduling, maps, and activity goals.
  Interventions: Behavioral: Implementation Intention Condition

INTERVENTIONS:
Behavioral: Control Group — Participants will wear a Fitbit Zip for 5 weeks to record their daily activity data. The first week of the study will provide a baseline measurement of activity. After this week, participants in this condition will begin receiving daily emails asking them to report their step count in a questionnaire. Participants in the control group will be matched with the intervention group for how much contact they have with the researcher.
  Arms: Control group
Behavioral: Implementation Intention Condition — Participants will wear a Fitbit Zip for 5 weeks to record their daily activity data. The first week of the study will provide a baseline measurement of activity. After this week, participants will be asked to increase their steps incrementally by 2,000 steps each week for the subsequent four weeks. To help achieve their step goals, they will receive maps of different routes near their home and/or work of varying distances and step counts. They will be asked to review their schedule for the next day and identify times when they could add steps into their schedules, and to record their daily step data in the daily questionnaire.
  Arms: Implementation Intention Condition

SUMMARY:
The study goal is to design an intervention utilizing implementation intentions to help participants prospectively plan and visualize ways to increase activity for the next day among working adults who do not currently exercise or use an activity monitor. Investigators will assess the level of and changes in physical activity, and how this relates to various individual factors that are related to exercise and health, including self-efficacy, control beliefs, and cognition.

DETAILED DESCRIPTION:
The 5-week study consists of a 1-week baseline, where participants are asked to wear a Fitbit to document the number of steps taken that day to establish an objective measurement of steps before the intervention began. In the intervention condition, after the baseline week, during weeks 2 to 5, this condition is prompted with an email each evening for four weeks to review their schedules for the following day and identify time slots where they could add activity. They are given instructions for providing a detailed calendar of appointments and open slots for the next day using a simple daily planner. The planning implementation intention manipulation involves recording specific information about when, where, and how they will add steps to their day. They are provided with maps near their home and work with specific information about distances, estimated time to walk between different points, and number of steps for specific routes to help them in planning for specific routes.The control condition is matched for how much contact they have with the research staff (called and emailed the same amount of times) and also wear the Fitbit daily. The only difference from the intervention group is that they do not get the daily planning instructions or maps for the implementation intention strategy treatment. All activity data from the Fitbit was deidentified and aggregated with an online platform called Fitabase.

ELIGIBILITY:
Inclusion Criteria:

* Currently working full time
* Not engaged in regular exercise
* 35 years of age or older

Exclusion Criteria:

* Not healthy enough to engage in a walking intervention

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margie Lachman, Ph.D., Principal Investigator — Brandeis University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson SA, Lachman ME. Perceived Control and Aging: A Mini-Review and Directions for Future Research. Gerontology. 2017;63(5):435-442. doi: 10.1159/000468540. Epub 2017 Apr 8. PMID 28391279
- [Background] Robinson, S. A. & Lachman, M. E. (2016). Perceived Control and Behavior Change: A Personalized Approach. In F. Infurna & J. Reich (Eds.), Perceived Control: Theory, Research, and Practice in the First 50 Years (pp. 201-227). New York, New York: Oxford University Press.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Implementation Intention Condition
Started (Number of participants enrolled in study and randomly assigned to group) | 32 | 31
Pre-test (Number of participants that filled out pre-test measures and started the study) | 30 | 30
Completed (Number of participants that completed the study) | 30 | 29
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Participants will wear a Fitbit Zip to record their daily activity data, which was deidentified and aggregated with an online platform called Fitabase. Participants in the control group will be matched with the intervention group for how much contact they have with the researcher.
  Participants will wear a Fitbit Zip for 5 weeks to record their daily activity data. The first week of the study will provide a baseline measurement of activity. After this week, participants in this condition will begin receiving daily emails asking them to report their step count in a questionnaire. Participants in the control group will be matched with the intervention group for how much contact they have with the researcher.
- Total: Total of all reporting groups
Arm/Group | Control Group | Implementation Intention Condition | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 30 | 59
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.22 (7.68) | 46.33 (8.03) | 49.37 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 32 | 31 | 63

OUTCOME MEASURES:

1. Primary Outcome: Steps
Description: Weekly average of daily step counts with Fitbit (averaged across 7 days at Week 1 and averaged across 7 days at Week 5).
Time Frame: Week 1 & Week 5
Population: Analysis population based on participants that successfully synced their Fitbit and did not withdraw before the start of the study.
Measure: Mean (Standard Deviation); unit: Daily Steps
Arm/Group | Control Group | Implementation Intention Condition
Number analyzed (Participants) | 30 | 30
Daily Steps
  Week 1 | 6337.77 (2207.44) | 6966.06 (2818.05)
  Week 5 | 6109.46 (3308.75) | 8900.35 (4416.04)
Statistical Analysis 1: Comparison: Control Group vs Implementation Intention Condition; Test type: Superiority; p = .006, Mixed Models Analysis; Controlling for age, gender, and functional health

2. Primary Outcome: Activity Intensity
Description: Weekly average of daily time spent in moderate to vigorous intensity activity (averaged across 7 days at Week 1 and averaged across 7 days at Week 5).
Time Frame: Week 1 & Week 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Control Group | Implementation Intention Condition
Number analyzed (Participants) | 30 | 30
Minutes
  Week 1 | 18.71 (20.31) | 22.25 (22.05)
  Week 5 | 18.51 (25.84) | 32.23 (30.73)
Statistical Analysis 1: Comparison: Control Group vs Implementation Intention Condition; Test type: Superiority; p = .034, Mixed Models Analysis; Controlling for age, gender, and functional health

3. Secondary Outcome: Cognitive Composite Score
Description: Z-score composite on the Brief Test of Adult Cognition by Telephone (BTACT). Individual tests scores were first standardized to z-scores. The z-score composite was calculated by averaging the z-scores of the 5 tests: word list immediate, word list delayed, backwards counting, digits backwards, and category fluency. Post-test z-scores were standardized based on the mean and s.d. of the pretest scores. A higher z-score is indicative of better cognitive functioning.
Time Frame: Baseline (Pre-Test) and Week 5 (Post-Test )
Population: Analysis population based on those who completed cognitive test at each testing point.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Control Group | Implementation Intention Condition
Number analyzed (Participants) | 30 | 30
Z-score
  Pre-Test | -.17 (.70) | .17 (.48)
  Post-Test | .21 (.50) | .65 (.52)
Statistical Analysis 1: Comparison: Control Group vs Implementation Intention Condition; Test type: Superiority; p = .065, Mixed Models Analysis; Controlling for age, gender, and education

4. Secondary Outcome: Exercise Control Beliefs
Description: Degree of perceived control over Exercise. Range from 1 (Strongly agree) to 5 (strongly agree). Reverse coded so that a higher number indicates more perceived control over exercise.
Time Frame: Baseline (Pre-Test) and Week 5 (Post-Test )
Population: Analysis population based on those who completed Control Beliefs over Exercise questionnaire at each testing point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Implementation Intention Condition
Number analyzed (Participants) | 28 | 23
units on a scale
  Pre-Test | 4.26 (.52) | 4.26 (.72)
  Post-Test | 4.32 (.54) | 3.90 (.85)
Statistical Analysis 1: Comparison: Control Group vs Implementation Intention Condition; Test type: Superiority; p = .308, Mixed Models Analysis; Controlling for age, gender, and level of education

5. Secondary Outcome: Exercise Self-efficacy
Description: Amount of confidence in ability to exercise.
Time Frame: Baseline (Pre-Test) and Week 5 (Post-Test )
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Implementation Intention Condition
Number analyzed (Participants) | 27 | 23
units on a scale
  Pre-test | 2.15 (0.99) | 2.19 (0.81)
  Post-test | 2.16 (0.86) | 2.29 (0.92)
Statistical Analysis 1: Comparison: Control Group vs Implementation Intention Condition; Test type: Superiority; p = .349, ANOVA

6. Secondary Outcome: Exercise Self-efficacy Beliefs - Time Composite
Description: Amount of confidence in ability to exercise when facing time constraints. Range from 1 (Very Sure) to 4 (Not sure at all). Reverse coded so that a higher number indicates more self-efficacy. 3 items, summed to form time-relevant composite scale.
Time Frame: Baseline (Pre-Test) and Week 5 (Post-Test )
Population: Analysis population based on those who completed Exercise Self-efficacy Beliefs questionnaire at each testing point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Implementation Intention Condition
Number analyzed (Participants) | 24 | 23
units on a scale
  Pre-Test | 1.96 (1.05) | 1.90 (.75)
  Post-Test | 1.94 (.89) | 2.30 (.90)
Statistical Analysis 1: Comparison: Control Group vs Implementation Intention Condition; Test type: Superiority; p = .022, Mixed Models Analysis; Controlling for age, gender, and level of education

ADVERSE EVENTS:
Groups:
- Control Group: Participants will wear a Fitbit Zip to record their daily activity data, which will be deidentified and aggregated with an online platform called Fitabase. Participants in the control group will be matched with the intervention group for how much contact they have with the researcher.
  Assigned Intervention - Participants will wear a Fitbit Zip for 5 weeks to record their daily activity data. The first week of the study will provide a baseline measurement of activity. After this week, participants in this condition will begin receiving daily emails asking them to report their step count in a questionnaire. Participants in the control group will be matched with the intervention group for how much contact they have with the researcher.
Arm/Group | Control Group | Implementation Intention Condition
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No